CLINICAL TRIAL: NCT04787432
Title: The Effect of Salutogenic Model Based Frailty Prevention Program on Development of Frailty and Sense of Coherence in Women Aged 55 Years and Over
Brief Title: Salutogenic Frailty Prevention Program for Women Aged 55 Years and Over
Acronym: SAFRAPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Merve ALTINER YAS, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IU-Cerrahpasa
Record Dates: First submitted 2021-03-02; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Frailty; Frailty Syndrome; Salutogenesis; Sense of Coherence
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Experimental: SAFRAPP Intervention
  Participants in this group will receive a 6-week SAFRAPP intervention, comprising of laughter yoga, health education and case management. SAFRAPP will be conducted on social media (Facebook and WhatsApp).
  Interventions: Behavioral: Salutogenic Frailty Prevention Program
- Control Grup (No Intervention): The control group will not receive any intervention during the study. Participants in the control group will take the same program after the study is completed.

INTERVENTIONS:
Behavioral: Salutogenic Frailty Prevention Program — Laughter yoga: The first component of intervention is the laughter yoga that is a combination of warm up exercise, deep breathing exercises, childlike playfulness and laughter exercises. Each session of laughter yoga will be offered twice a weekly and 40 minutes each time.
  Health education: The second component of intervention consisted of six health issues which are "health, frailty and generalized sources of resistance for frailty", the most common medical condition and medication use", "physical activity", "healthy diet", "falls prevention" and "cognitive and psychosocial well-being".
  Case management: The third component of intervention is activities that determine each participant's health needs with the Omaha System and support them for the use of appropriate resources.
  Arms: Intervention

SUMMARY:
Frailty is a condition of reduced the capacity in multiple body systems and causing adverse outcomes because of decreasing the ability to cope with stressors. Female sex, the changes of the body imposed by ageing, and coping strategies for stressors are causal mechanisms in the development of frailty. This project is designed with the salutogenic model that is focused on the concepts of health, stress, and coping. The aim of this project is to assess the effect of Salutogenic Frailty Prevention Program on promoting sense of coherence and preventing the development of frailty in women aged 55 years and over

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study
* Woman aged 55 years and over
* Pre-frail (Total FRAIL scale score 1 or 2)
* Has Internet access

Exclusion Criteria:

* To be semi-dependent and dependent according to the Katz Daily Activities Activity Scale
* To have any cognitive, psychiatric and neurological disorders
* To have any surgical operation in the past 3 month
* Communication barrier (due to hearing/vision impairment)

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change in Sense of Coherence | Baseline, 3 months, 6 months, 9 months
  Sense of coherence assesses an individual's orientation and internal strengths. It consists of 13 items rated on a 7-point Likert scale, and has three components including comprehensibility (5-item), manageability (4-item) and meaningfulness (4-item)
Change in FRAIL scale | Baseline, 3 months, 6 months, 9 months
  The FRAIL scale consists of 5 items (fatigue, resistance, ambulation, illnesses, loss of weight). Frail scale scores range from 0-5 and represent frailty status as frail (3-5), pre-frail (1-2), and robust (0).

SECONDARY OUTCOMES:
Change in The World Health Organisation- Five Well-Being Index (WHO-5) | Baseline, 3 months, 6 months, 9 months
  The five-items Well-Being Index will be used to assess participants' psychological well-being.
Change in health-related quality of life | Baseline, 3 months, 6 months, 9 months
  The EQ-5D-3L descriptive system evaluates the participants' health state in the five dimensions including mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Change in EQ-VAS | Baseline, 3 months, 6 months, 9 months
  EQ visual analogue scale (EQ-VAS) is a vertical scale that assesses the participant's own judgement regarding their health between 0 and 100.
Change in number of falls | Baseline, 3 months, 6 months, 9 months
  Participants will be asked about the number of falls in the past three months
Change in fear of fall | Baseline, 3 months, 6 months, 9 months
  Participants will be asked a single question: Are you afraid of falling? The possible answers were never afraid," sometimes afraid," afraid, and always afraid.
Change in number of emergency admissions | Baseline, 3 months, 6 months, 9 months
  Participants will be asked about the number of the emergency visit in the past 3 months

REFERENCES:
- [Derived] Yas MA, Secginli S. Salutogenic Model-Based Frailty Prevention Program for Pre-Frail Women Aged 55 Years and Over (SAFRAPP): A Study Protocol for a Randomized Controlled Trial. Res Theory Nurs Pract. 2022 Apr 1;36(2):215-232. doi: 10.1891/RTNP-2021-0098. PMID 35584890